CLINICAL TRIAL: NCT00135057
Title: Insulin Glulisine Administered in a Fixed Bolus Regimen Versus Variable Bolus Regimen Based on Carbohydrate Counting in Adult Subjects With Type 2 Diabetes Receiving Insulin Glargine as Basal Insulin
Brief Title: Insulin Glulisine in Adult Subjects With Type 2 Diabetes Receiving Insulin Glargine as Basal Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_3502
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin glulisine; Insulin Glargine

INTERVENTIONS:
Drug: insulin glulisine
Drug: insulin glargine

SUMMARY:
The purpose of this study is to compare the change in glycemic control, as measured by hemoglobin A1c (HbA1c) from baseline to study week 24, in subjects receiving insulin glulisine as mealtime insulin following a variable bolus insulin regimen (based on carbohydrate counting) versus a fixed bolus insulin regimen, with insulin glargine as basal insulin in both arms of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus for at least six months; 18 to 70 years of age, inclusive.
* A1c ≥ 7.0% and ≤ 10% at screening
* At least 3 months of continuous insulin and/or insulin analogue therapy (on at least 2 injections) +/- metformin prior to study entry. (Note: Subjects receiving insulin glargine [Lantus] twice a day [split dose] will be considered as being on one injection only.)
* Willingness of subject to discontinue other anti-diabetic drug treatments and to remain off them through the entire study
* Negative glutamic acid decarboxylase (GAD) autoantibodies
* Ability and willingness to perform self-monitoring of blood glucose (SMBG) at least four times a day, and at least 7 times daily during the 7-point blood glucose (BG) profile measurement days
* Ability and willingness to adhere to, and be compliant with, the study protocol
* Must be able to read English at the sixth grade level in order to complete the patient-reported outcomes component of the study.
* Signed informed consent

Exclusion Criteria:

* Subjects treated with sulfonylureas, thiazolidinediones (TZDs), or any other oral antidiabetic drugs (within the 3 months before study entry) except for insulin and/or insulin analogues with or without metformin
* Planned pregnancy; or pregnant or lactating females.
* For subjects treated with metformin: serum creatinine ≥ 1.5 mg/dL (133 µmol/L) for males or ≥ 1.4 mg/dL (124 µmoL) for females
* Serum creatinine ≥ 3.0 mg/dL (266 µmol/L)
* Any clinically significant renal disease (other than proteinuria) or hepatic disease
* Serum ALT or AST levels greater than 2.5 X the upper limit of normal
* Any current malignancy or any cancer within the past 5 years (except for adequately treated basal cell skin cancer or cervical carcinoma in situ)
* Diagnosis of dementia or mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Diagnosis of impaired dexterity or vision rendering the subject unable to administer multiple daily injections (MDIs)
* Cardiac status New York Heart Association (NYHA) III-IV
* Hypersensitivity to Lantus or insulin glulisine (Apidra) or any of their components
* Any disease or condition (including abuse of illicit drugs, prescription medicines or alcohol) that, in the opinion of the investigator or sponsor, may interfere with the completion of the study.
* Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281
Dates: Start 2004-04; Study Completion 2005-08

PRIMARY OUTCOMES:
Compare the change in glycemic control (as measured by A1c) from baseline to endpoint of fixed dose bolus regimen vs. variable bolus regimen based on carbohydrate count

CONTACTS AND LOCATIONS:
Overall Officials: Karen Barch, B.S., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States

REFERENCES:
- [Derived] Bergenstal RM, Johnson M, Powers MA, Wynne A, Vlajnic A, Hollander P, Rendell M. Adjust to target in type 2 diabetes: comparison of a simple algorithm with carbohydrate counting for adjustment of mealtime insulin glulisine. Diabetes Care. 2008 Jul;31(7):1305-10. doi: 10.2337/dc07-2137. Epub 2008 Mar 25. PMID 18364392